CLINICAL TRIAL: NCT06209385
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of YZJ-5053 Tablets in Participants With Advanced Solid Tumors
Brief Title: A Phase 1 Study of YZJ-5053 Tablets in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-5053-1-01
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YZJ-5053 tablets (Experimental): YZJ-5053 tablets will be administrated orally quaque die (QD) for 21 days
  Interventions: Drug: YZJ-5053 tablets

INTERVENTIONS:
Drug: YZJ-5053 tablets — YZJ-5053 tablets will be administrated orally QD for 21 days
  Other Names: SHY-1901

SUMMARY:
The goal of this study is to evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of YZJ-5053 Tablets in Participants with Advanced Solid Tumors

DETAILED DESCRIPTION:
Part1(phase 1a) :To define the maximum tolerated dose (MTD) and/or a recommended phase 2 dose(RP2D). To evaluate the safety and tolerability of YZJ-5053 tables in participants with advanced solid tumors.

Part2(phase 1b) : To define the RP2D. To evaluate the safety and tolerability of YZJ-5053 tables in subjects with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects are ≥ 18 years of age on the day of signing the informed consent.
* Histologically or cytologically confirmed advanced or metastatic solid tumors who have failed standard treatment, or are ineligible for the standard treatment, or have no standard treatment, or declined standard treatment.
* Subjects must have at least one measurable target lesion in indication expansion phase (Part 2) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria which has not received radiotherapy (or progressive disease after radiotherapy), or at least one evaluable lesion in dose escalation phase (Part 1) .
* Subjects with previously confirmed brain metastases were enrolled if they were clinically asymptomatic, in stable condition, and did not require steroid therapy for at least 4 weeks before the initiation of study treatment.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1;
* Life expectancy at least 3 months;
* Adequate hematologic and organ function at screening and within 28 days prior to initiation of study treatment (without receiving any blood transfusion or hematopoietic stimulating factors within 2 weeks prior to screening),as evidenced by:

absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L； Platelets ≥ 75 x 10^9/L； Hemoglobin ≥85 g/L； aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) , or ≤ 5 x ULN if liver cancer or liver metastases are present.

Total bilirubin < 1.5 x ULN , or < 3.0 x ULN for subjects with liver cancer or liver metastases or documented Gilbert's syndrome (unconjugated hyperbilirubinemia)； Serum creatinine (Scr) <1.5×ULN, or creatinine clearance (Ccr) > 50 mL/min according to Cockcroft-Gault equation; international normalized ratio (INR) and activated partial thromboplastin time (APTT) < 1.5 ULN;

* A woman of child-bearing potential (WOCBP) must have a negative serum pregnancy test prior to initiation of study treatment (serum pregnancy test is not required for females of nonchild-bearing potential who have undergone surgical sterilization, such as hysterectomy and/or bilateral oophorectomy, or those who have not experienced menses for 12 consecutive months and are judged to be postmenopausal based on factors such as age and castration therapy).
* Subjects must agree to use adequate contraceptive methods prior to initiation of study treatment, during the study, and for at least 28 days following the last dose of YZJ-5053 tablets.

Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding.
* History of malignancy within 3 years prior to screening, with the exception of the cancer under investigation in this study and curatively treated carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer or any other tumor that has been treated curatively and with no evidence of disease for at least 3 years (for indication expansion phase [1b] only).
* Presence of uncontrolled pleural effusion, pericardial effusion, or ascites that require recurrent drainage procedures (monthly or more frequently).
* Impaired cardiac function or clinically significant cardiovascular disease.
* Conditions or diseases that impair gastrointestinal (GI) function which may significantly alter the absorption of YZJ-5053 tables (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Subjects with active infection requiring intravenous (IV) antibiotics at the time of screening or within 2 weeks prior to initiation of study treatment.
* Subjects with positive HIV antibody, or positive hepatitis B surface antigen (HBsAg) with hepatitis B virus (HBV) DNA ≥2×10^3 IU/ml (equivalent to 10^4 copies/ml), or positive hepatitis C virus antibody at the time of screening;
* Have received chemotherapy within 3 weeks, and radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy or any other anti-tumor therapy within 4 weeks prior to initiation of study treatment.
* Subject who could not discontinue use of strong inhibitors or strong inducers of Cytochrome P450 3A (CYP3A) and Cytochrome P450 2C8 (CPY2C8) during the study period.
* Subjects who have received a live vaccine or live attenuated vaccine within 4 weeks prior to initiation of study treatment.
* Subjects who have previously received adenosine A2a receptor (A2aR) antagonists or A2aR/adenosine A2b receptor (A2bR) antagonists.
* Adverse events (AEs) from previous antitumor therapy have not recovered to baseline or to CTCAE Grade 1 prior to initiation of study treatment, excluding subjects with alopecia (any grade), peripheral sensory neuropathy (Grade ≤ 2), and any other toxicities of no clinical significance (Grade ≤ 2);
* Subjects with a known history of autoimmune thyroid disease such as diffuse toxic goiter (Graves disease) , acute or subacute thyroiditis. Subjects with active autoimmune diseases or a known history of autoimmune diseases that potentially relapsing, exception:

Subjects with autoimmune-related hypothyroidism requiring stable dose thyroxine replacement only are eligible; Subjects with type I diabetes mellitus controlled on a stable insulin regimen are eligible;

* Subjects who have received systemic corticosteroids (> 10 mg/day prednisone equivalent) or other systemic immunosuppressants (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs) within 4 weeks prior to the initiation of study treatment, but excluded:

Locally, ocularly, intra-articularly, intranasally, or inhaled corticosteroids; Subjects receiving acute low-dose systemic immunosuppressive drugs (e.g., single dexamethasone for nausea) may be enrolled after discussion with and approval from medical monitor ; Alternative steroid doses for diseases such as adrenal or pituitary insufficiency are ≤ 10 mg/day in prednisone equivalents; Corticosteroids hydrochloride (eg fludrocortisone) for orthostatic hypotension; Short-term (≤ 7 days) use of steroids for the prevention or treatment of non-autoimmune allergic diseases; Single ues of glucocorticoids before enhanced-imaging for prevention of contrast agent allergy;

* Major surgical procedures, within 4 weeks prior to initiation of study treatment, or anticipation of need for major surgical procedure during the study period.
* Other severe and/or uncontrolled concomitant medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol.
* Presence of other conditions, therapy, or laboratory abnormalities that, in the opinion of the investigator, might confound the results of the study and interfere with the subject's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) of YZJ-5053 | 21days as a cycle
  The MTD will be based on dose limiting toxicity (DLT)
To identify a recommended Phase 2 dose (RP2D) of YZJ-5053 | 21days as a cycle
  RP2D will be be based on MTD
Number of participants with treatment-related adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) | 21days as a cycle
  All events with a Grade 3 or above toxicity (defined by the NCI-CTCAE 5.0) will be tabulated by event and by relationship to YZJ-5053

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  Maximum plasma concentration of YZJ-5053 after single and multiple dose administration of YZJ-5053
Time to reach Cmax (Tmax) of YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  The amount of time to reach Cmax after single and multiple dose administration of YZJ-5053
Terminal half-life (t1/2) of YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  Terminal half-life (t1/2) after single and multiple dose administration of YZJ-5053
Area under the plasma concentration-time curve (AUC) of YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  Area under the plasma concentration versus time curve after single and multiple dose administration of YZJ-5053
apparent clearance following oral administration for YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  To characterise the pharmacokinetics (PK) after single and multiple dose administration of YZJ-5053
apparent volume of distribution for YZJ-5053 | single dose: predose, 0.5、1、2、4、6、8、12、24、48、72 hours post-dose. multiple dose: predose on days 1、3、4、5、6, and 0.5、1、2、4、6、8、12 hours post-dose on day 5
  To characterise the PK after single and multiple dose administration of YZJ-5053
Objective Response Rate (ORR) as defined by Investigator-assessed Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Evaluate every 6 weeks (±1 week) until study completion, an average of 1 year
  For solid tumors, this will be determined per RECIST v1.1 guidelines
Disease control rate (DCR) as defined by Investigator-assessed RECIST v1.1 | Evaluate every 6 weeks (±1 week) until study completion, an average of 1 year
  For solid tumors, this will be determined per RECIST v1.1 guidelines
Duration Of Response (DOR) as defined by Investigator-assessed RECIST v1.1 | Evaluate every 6 weeks (±1 week) until study completion, an average of 1 year
  For solid tumors, this will be determined per RECIST v1.1 guidelines
Progression-free Survival (PFS) as defined by Investigator-assessed RECIST v1.1 | Evaluate every 6 weeks (±1 week) until study completion, an average of 1 year
  For solid tumors, this will be determined per RECIST v1.1 guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital
Locations (4):
- China (4):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No